CLINICAL TRIAL: NCT02554175
Title: The Effective Effect-Site Propofol Concentration for Induction and Intubation for Schnider Model in Parturients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Tingting Wang, Obstetrics and Gynecology Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTWang
Record Dates: First submitted 2015-08-26; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: C.Delivery; Surgery (Previous), Gynecological
Keywords: Propofol; Schnider model
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- the target propofol concentration (Experimental): patients were allocated to 1 of 6 groups of predefined propofol target Ce for induction, namely, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5 µg.mL-1.Propofol was administered to achieve target propofol Ce.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol was administered to achieve target propofol Ce

SUMMARY:
The aim of this study was to determine the target propofol concentration needed to provide adequate hypnosis for induction and tracheal intubation for Schnider model using total body weight (TBW) in parturients. In addition, investigators wanted to define the hemodynamic adverse effects associated with these propofol target concentrations.

DETAILED DESCRIPTION:
The temperature was maintained at 22˚ C in the operating room. Patients were placed supine with 15°left lateral tilt achieved using a wedge under the right buttock. Electrocardiograph (ECG), pulse oxygen saturation (SpO2), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and heart rate (HR) were monitored by one anesthesiologist (S/5 Anesthesia Monitor, GE Healthcare, Helsinki, Finland), and Bispectral Index (BIS) values (A2000 BIS® XP monitor, version 3.2; Aspect Medical Systems Inc., Newton, MA) were obtained and recorded. The BIS smoothing time period was set at 15 seconds. The mean values of the above-mentioned parameters were recorded at 3-min intervals for three consecutive times to determine baseline values. Peripheral vein catheterization on the right hand was then performed but no prehydration was given. A fixed volume of 500 mL hydroxyethyl starch solution was infused at the rate of 0.2 ml.kg-1.min-1, then Lactated Ringer's solution was infused at the same rate until the end of surgery.

Using a computer-generated random-number sequence, patients were allocated to 1 of 6 groups of predefined propofol target Ce for induction, namely, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5 µg.mL-1. General anesthesia was induced with fentanyl 3 µg.kg-1. Propofol was administered by the TCI device to achieve the predetermined target propofol Ce. Loss of consciousness was defined by the disappearance of the eyelash reflex that was assessed every 5 seconds after patients spontaneously closed their eyes. After loss of consciousness, succinylcholine 1.5 mg.kg-1 was administered and tracheal intubation was performed 1 minutes later only if the BIS value was <60 and target propofol Ce had been reached. After intubation, patients were connected to mechanical ventilation adjusted to obtain an end-tidal CO2 of 30 to 35 mm Hg and the propofol target concentration was reduced to 3µg.mL-1. Anesthesiologists performing loss of consciousness assessment and intubation were blinded to the target propofol Ce. SpO2, SBP, DBP, MAP and HR were recorded once a minute for 10 min until 5 minutes after tracheal intubation when the study finished.

ELIGIBILITY:
Inclusion Criteria:

* Thirty-six women undergoing elective cesarean section under general anesthesia were enrolled in this prospective observational study.

Exclusion Criteria:

* Diabetes controlled by insulin
* Preeclampsia
* Heart diseases
* History of taking drugs potentially affecting cardiovascular system.
* Patients fasted for at least 8 hours before surgery and no premedication was given

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
target propofol concentration needed to provide adequate hypnosis for induction and tracheal intubation for Schnider model using total body weight (TBW) in parturients | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaoqiang Huang, Study Director — Department of Anesthesiology, Obstetrics and Gynecology Hospital of Fudan University, Shanghai, China